CLINICAL TRIAL: NCT00951171
Title: Evaluation of the Effect of Cervical Occlusion During Infertility Treatment by Intrauterine Insemination
Brief Title: Effect of Cervical Occlusion During Intrauterine Insemination (IUI)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Randomization flawed. Results were poor in the innovative catheter group
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Andrew Blazar, M.D., Prinicpal Investigator, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO_IUI
Record Dates: First submitted 2009-07-31; First posted 2009-08-04 (Estimated); Results first posted 2012-08-28 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cervical occulsion (Experimental): Insemination Eliptosphere catheter filled with 1cc of air for 15 minutes. H/S Eliptosphere by Copper surgical (U.S. Patent No. 5,624,399)
  Interventions: Procedure: Intrauterine Insemination
- Standard IUI (Active Comparator): Insemination with TOmcat catheter
  Interventions: Procedure: IUI with the standard inseminator

INTERVENTIONS:
Procedure: Intrauterine Insemination — The intervention arm will undergo temporary (15 minutes) cervical occlusion with the eliptosphere intracervical catheter. This catheter is typically used to perform saline infusion ultrasounds to image the uterine cavity in our practice.
  Other Names: H/SH
  Arms: Cervical occulsion
Procedure: IUI with the standard inseminator — The control arm will undergo insemination with the standard inseminator (TOmcat catheter).
  Arms: Standard IUI

SUMMARY:
Study Hypothesis: There is a difference in pregnancy rates between intrauterine insemination (IUI) in cycles performed with cervical occlusion by a balloon catheter designed for sonohysterograms as compared to those performed with a standard inseminator.

The investigators will compare pregnancy rates in patients undergoing routine IUI either with balloon occlusion or with standard insemination. The patients will receive the standard clinical care per the investigators' office guidelines, except they will be randomized to insemination with either of two catheters.

DETAILED DESCRIPTION:
An open speculum will be used and patients will undergo insemination with their partners sperm (same quantity in both arms). If randomized to treatment arm a balloon catheter will be filled with 1cc of air prior to insemination. The speculum will be removed immediately and the catheter will be left in for 15 minutes and then removed. Pregnancy outcomes will be recorded in both groups.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing IUI for unexplained infertility in our office: Center for Reproduction and Infertility (Providence, RI)

Exclusion Criteria:

* "Abnormal" Semenalysis TMC < 5 million
* Blocked Fallopian tubes

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2009-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Blazar, MD, Principal Investigator — Women & Infants Hospital
Locations (1):
- Center for Reproduction and Infertility, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients recruited were women scheduled previously for IUI for treatment of unexplained infertility at the WIHRI office.
Pre-assignment Details: 2 patients in the occlusion group experienced pain and were immediately transferrred to the standard group,thereby creating an apparent discrepancy in numbers
Period: Overall Study
Arm/Group | Cervical Occulsion | Standard IUI
Started | 40 | 55
Pregnancy | 1 | 7
Completed | 38 | 55 (2 of the cervical occlusion group transferred to standard group because of pain during attempted IUI)
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervical Occulsion | Standard IUI | Total
Number analyzed (Participants) | 40 | 55 | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 55 | 95
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 55 | 95
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 55 | 95

OUTCOME MEASURES:

1. Primary Outcome: Clinical Pregnancy
Description: positive beta HCG test
Time Frame: 1 month
Population: All study women undergoing IUI were included
Measure: Number; unit: positive pregnancy test (beta HCG)
Arm/Group | Cervical Occulsion | Standard IUI
Number analyzed (Participants) | 40 | 53
positive pregnancy test (beta HCG) | 1 | 7

2. Secondary Outcome: Live Birth
Time Frame: 9 months
Reporting Status: Not Posted

3. Secondary Outcome: Positive Pregnancy Test
Time Frame: 14 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Cervical Occulsion | Standard IUI
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/55
Other Adverse Events (participants affected / at risk) | 2/40 | 0/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cervical Occulsion (N=40) | Standard IUI (N=55)
pain with device (Surgical and medical procedures) | 2/2 (2) | 0/0 (0)

LIMITATIONS AND CAVEATS:
Randomization method found to be faulty

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes